CLINICAL TRIAL: NCT02495441
Title: A Comparison of Rapid Immunoassay Tests for the Detection of Ruptured Membranes
Brief Title: Rapid Immunoassay Tests for the Detection of Ruptured Membranes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: De Soysa Hospital for Women (Other)
Collaborators: Clinical Innovations, LLC (Industry)
Responsible Party: Principal Investigator, Hemantha M. Senanayake, Professor of Obstetrics and Gynecology, De Soysa Hospital for Women
Other Study IDs: PROM
Record Dates: First submitted 2015-07-01; First posted 2015-07-13 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Premature Rupture of Membranes
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dribbling group: Any woman who presents with alleged leakage of amniotic fluid. They will under go rapid Immunoassay Tests for the Detection of PROM
  Interventions: Other: Use of Rapid Immunoassay Tests for the Detection of PROM

INTERVENTIONS:
Other: Use of Rapid Immunoassay Tests for the Detection of PROM — After informed consent , both the ROM Plus®, ActimProm Amnioquick® Complete and AmniSure® bedside tests (without the use of a speculum) will be performed.
  The patient will then undergo the standard clinical assessment, which includes a sterile speculum exam (SSE). If either 1) amniotic fluid is seen leaking from the cervical os, or 2) if at least two of the following three clinical signs are present: visual pooling of fluid in the posterior fornix, positive nitrazine test, and microscopic evidence of ferning, then the patient will be considered positive for ROM.
  Women who cannot be confirmed clinically by the SSE will undergo an ultrasound evaluation to determine the amniotic fluid index. The patient will be treated according to the results of the SSE and ultrasound, not the results of IGFBP-1/AFP tests and Amnisure®.

SUMMARY:
The aim of the study is to demonstrate substantial equivalence of IGFBP-1/AFP tests with the "predicate device" Amnisure® in detecting pre labor rupture of membranes. 4 test kits are compared against a common referent standard (gold standard), which is clinical assessment.

DETAILED DESCRIPTION:
Premature rupture of membranes (PROM) is defined as spontaneous rupture of membranes (ROM) before the onset of uterine contractions. Its diagnosis is often obvious with the woman presenting with leakage of amniotic fluid, but it could also turn out to be a difficult diagnostic dilemma.

The diagnosis of fetal membrane rupture is conventionally made using a clinical assessment. First, by speculum examination, the clinician looks for amniotic fluid leaking from the cervical os. If clear fluid is visualized leaking from the cervical os, the diagnosis is positive for fetal membrane rupture. More commonly, leaking is absent, and a more extensive workup is required, which includes nitrazine/pH testing, visual inspection of pooling of fluid in the posterior fornix, and a microscopic evaluation of the collected specimen (ferning). Although this approach is considered the standard of care, it is fraught with inaccuracies, requires an intrusive examination and may not provide a rapid diagnosis.

Rapid, point of care, qualitative immunochromatographic tests (ie., Amnisure®, ActimProm®, Amnioquick® Complete and ROM Plus®) that detect proteins found in amniotic fluid at high concentrations, have been used to diagnose the rupture of membranes (ROM) for several years. In many hospitals, Amnisure® has replaced the sterile speculum exam as the standard of care for diagnosing ROM. It identifies Placental Alpha Microglobulin-1 (PAMG-1), a 34 kd fetal glycoprotein, in cervicovaginal secretions.

ROM Plus® ActimProm®and Amnioquick® Complete+ are newer additions into the market for testing for PROM. Both these tests use a monoclonal/polyclonal antibody approach to detect two different proteins found in amniotic fluid at high concentrations. They detect Placental Protein-12 (also known as Insulin-like Growth Factor Binding Protein-1 - IGFBP-1) as well as Alpha Fetoprotein (AFP).

The aim of the study is to demonstrate substantial equivalence of IGFBP-1/AFP tests with the "predicate device" Amnisure®. Stated in statistical terms, the aim is to demonstrated that IGFBP-1/AFP tests are non-inferior to Amnisure® in terms of sensitivity and specificity when both are compared in a paired-sample fashion to a common referent standard (gold standard), which is clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Any woman who presents with alleged leakage of amniotic fluid is eligible for recruitment

Exclusion Criteria:

* Known placental previa
* Active vaginal bleeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes the pregnant mothers presenting to the De Soysa Hospital for Women, Colombo with alleged leakage of amniotic fluid. This is an urban population with multiple ethical back grounds.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants that become positive for pre labor rupture of membranes by the immunological test kits. | up to 1 year
  This will be assessed by the performing 4 immunological tests and clinical assessment. These test kits includes ROM Plus, ActimProm®, Amnioquick® and Amnisure. Outcomes of the immune tests will be compared against a gold stranded clinical assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Hemantha Senanayake, MS, FRCOG, Principal Investigator — Department of Obstetrics & Gynaecology Faculty of Medicine University of Colombo, Sri Lanka
Locations (1):
- De Soyza Hospital for Women, Colombo, Western Province, Sri Lanka